CLINICAL TRIAL: NCT00032708
Title: A Double Blind, Randomized Dose Response Study of Dryvax Vaccine Against Smallpox in Previously Vaccinated Adults
Brief Title: Dryvax Dilution-Prev Vacc Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01-651
Record Dates: First submitted 2002-03-28; First posted 2002-03-29 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-05

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — Smallpox Vaccine

INTERVENTIONS:
Biological: Dryvax

SUMMARY:
A double-blind, randomized, dose-response study of four dilutions of Dryvax in previously vaccinated adults in order to assess the clinical success rates, humoral responses, and virus-specific actifity of cytotoxi T cells and interferon-y producing T cells

ELIGIBILITY:
Inclusion Criteria:

* For cohort E (never vaccinated): Aged 18-31; Never been vaccinated for smallpox.
* If female, not pregnant or lactating.
* Promise to use an effective method of birth control for 7 months after vaccination.
* Negative result on a test for HIV, AIDS, Hepatitis B and C.
* Acceptable as blood donors.
* For cohorts A, B, C, D (previously vaccinated): Aged 32 to 60 years; known history of smallpox vaccination with a typical vaccinia scar; no smallpox vaccination after 1971.
* Healthy adults (aged 18-60).

Exclusion Criteria:

* Eczema or history of eczema, or other chronic skin disorder.
* Pregnancy or lactation.
* History of immunodeficiency, liver disease, severe kidney impairment, malignancy, HIV, Hepatitis B, or Hepatitis C.
* Household contact with persons who are under 12 months of age, pregnant or lactating, or have any of the specified diseases.

Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2004-04; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University Health Sciences Center, St Louis, Missouri, United States